CLINICAL TRIAL: NCT05984238
Title: Endoscopic Application of Pulsed Electric Fields Using by the Endogenex Generation 2 ReCET System for Duodenal Mucosal Regeneration for EliMination of INsulin in the treatmENT of Type 2 Diabetes: a Randomized Double-blind Sham Controlled Trial to Evaluate Safety, Feasibility and Efficacy Study
Brief Title: A Trial to Evaluate Safety, Feasibility and Efficacy of the ReCET Procedure (EMINENT-2)
Acronym: EMINENT-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Endogenex (Unknown)
Responsible Party: Principal Investigator, Jacques J.G.H.M. Bergman, prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL83266.000.22
Record Dates: First submitted 2023-07-11; First posted 2023-08-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Duodenal ablation; Endoscopy; Electroporation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: This study is a single-center, double-blind, sham-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this study, both the study team and the study subjects are blinded to the treatment through the 24 week follow-up visit. While the endoscopist is not blinded to individual treatments, he or she is blinded to cohort level data and is not responsible for patient follow-up. At the 24 week visit, the subject and study team are unblinded. The subjects who received the sham treatment undergo ReCET.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- ReCET procedure (Active Comparator): Patients receive ReCET (Re-Cellularization via Electroporation Therapy), which is performed using the ReCET device.
  After which a 2 week isocaloric diet is followed, and then semaglutide, a GLP-1 receptor agonist is started.
  Interventions: Device: ReCET; Drug: Semaglutide, 1.0 mg/mL
- Sham procedure (Sham Comparator): Patients receive sham procedure, this consists of placing an Endogenex catheter, or a catheter with a similar circumference at the endoscopists discretion in the stomach and leaving it in place for 30 minutes.
  After which a 2 week isocaloric diet is followed, and then semaglutide, a GLP-1 receptor agonist is started
  Interventions: Drug: Semaglutide, 1.0 mg/mL; Other: Sham procedure

INTERVENTIONS:
Device: ReCET — Investigational product.
  Arms: ReCET procedure
Drug: Semaglutide, 1.0 mg/mL — Already registered medicine for type 2 diabetes
Other: Sham procedure — The sham control for the ReCET procedure.
  Arms: Sham procedure

SUMMARY:
The objective of this study is to evaluate the safety, feasibility and efficacy of pulsed electric field induced duodenal mucosal regeneration (ReCET system by the Endogenex with the Gen-2 catheter) combined with a GLP-1 receptor agonist (Semaglutide, Ozempic) in subjects with insulin-dependent type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety, feasibility and efficacy of pulsed electric field induced duodenal mucosal regeneration (ReCET system by the Endogenex with the Gen-2 catheter) combined with a GLP-1 receptor agonist (Semaglutide, Ozempic) in subjects with insulin-dependent type 2 diabetes mellitus and an adequate beta cell reserve in a randomized sham-controlled study. The aimed effect is an adequate or improved glucose regulation without the need for insulin therapy. Secondary effects include improved cardiovascular, hepatic, and metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes mellitus
2. 28 - 75 years of age
3. On daily long acting insulin dose ≤ 1 U/kg, with a stable dose (within 10%) over 1 month
4. BMI ≥ 24 and ≤ 42 kg/m2
5. HbA1c ≤ 64 mmol/mol (8.0%)
6. Fasting C-peptide ≥ 0.2 nmol/L (0.6 ng/ml)
7. Willing to comply with study requirements and able to understand and comply with signed informed consent

Exclusion Criteria:

1. Diagnosed with Type 1 Diabetes or with a history of ketoacidosis
2. Current use of multiple daily doses insulin or insulin pump.
3. Current or within the last 3 months use of a GLP-1 analogue.
4. Known autoimmune disease, as evidenced by a positive Anti-GAD test, including Celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
5. Previous GI surgery that could affect the ability to treat the duodenum such as subjects who have had a Bilroth 2, Roux-en-Y gastric bypass, or other similar procedures or conditions
6. History of chronic or acute pancreatitis
7. Known active hepatitis or active liver disease
8. Symptomatic gallstones or kidney stones, acute cholecystitis or history of duodenal inflammatory diseases including Crohn's Disease and Celiac Disease
9. History of coagulopathy, upper gastro-intestinal bleeding conditions such as ulcers, gastric varices, strictures, congenital or acquired intestinal telangiectasia
10. Use of anticoagulation therapy (such as phenprocoumon and acenocoumarol) which cannot be discontinued for 3-5 days before and 48 hours after the procedure and novel oral anticoagulants (such as rivaroxaban, apixaban, edoxaban and dabigatran) which cannot be discontinued for 48 hours before and 48 hours after the procedure in accordance with the local protocol
11. Use of P2Y12 inhibitors (clopidogrel, pasugrel, ticagrelor) which cannot be discontinued for 5 days before and 48 hours after the procedure in accordance with the local protocol. Use of aspirin is allowed.
12. Unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during treatment through 4 weeks post procedure phase
13. Taking corticosteroids or drugs known to affect GI motility (e.g. Metoclopramide)
14. Receiving weight loss medications such as Meridia, Xenical, or over the counter weight loss medications
15. Anemia, defined as Hgb < 6.2 mmol/l
16. Known history of severe permanent cardiac arrhythmia's with clinical symptoms
17. Significant cardiovascular disease, including known history of valvular disease or myocardial infarction, heart failure, transient ischemic attack, or stroke within 6 months prior to the screening visit
18. With any implanted electronic devices or duodenal metallic implants
19. eGFR or MDRD < 30 ml/min/1.73m^2
20. Active systemic infection
21. Active malignancy within the last 5 years
22. Not potential candidates for surgery or general anesthesia
23. Active illicit substance abuse or alcoholism
24. Pregnancy or wish getting pregnant in next year
25. Participating in another ongoing clinical trial of an investigational drug or device that can interfere with the current study.
26. Any other mental or physical condition which, in the opinion of the Investigator, makes the subject a poor candidate for clinical trial participation

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of procedure-related SAEs, UADEs, SADEs, AESIs [safety] | 24 weeks
  The incidence rate of procedure-related SAEs, UADEs, SADEs, AESIs 24 weeks post ReCET procedure.
Percentage of patients off insulin at 24 weeks [efficacy] | 24 weeks
  Percentage of patients free of insulin at 24 weeks post ReCET with an HbA1c ≤ 58 mmol/mol compared to sham.

SECONDARY OUTCOMES:
Secondary safety endpoint 1 - hypoglycemic events | Through study completion (1 to 1,5 year)
  Number of hypoglycemic events
Secondary safety endpoint 2 - SAEs | Through study completion (1 to 1,5 year)
  All SAEs
Secondary feasibility endpoint 1 - technical success rate | 24 weeks (after cross-over)
  Technical success rate, defined as percentage of subjects successfully completed the ReCET procedure (defined as ≥ 3 ablations).
Secondary feasibility endpoint 2 - GLP-1RA tolerability | Through study completion (1 to 1,5 year)
  Percentage of subjects adequately using and tolerating GLP-1RA (semaglutide).
Secondary efficay endpoint 1 - HbA1c 48 weeks | at 48 weeks
  Protocol driven number of subjects free of insulin at 48 weeks, including an HbA1c ≤ 58 mmol/mol.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques JG Bergman, MD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Busch CBE, van den Hoek K, Neefjes-Borst EA, Nieuwdorp M, van Baar ACG, Bergman JJHGM. Optimizing duodenal tissue acquisition for mechanistic studies of duodenal ablation in type 2 diabetes. Endosc Int Open. 2025 Jan 29;13:a25032135. doi: 10.1055/a-2503-2135. eCollection 2025. PMID 40007651
- See also: Website for people that are interested in participating. — https://onderzoekdiabetes.nl/